CLINICAL TRIAL: NCT02614170
Title: A Prospective Collection of Peripheral Blood and Urine Specimens to Study C-peptide and Insulin in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-115
Record Dates: First submitted 2015-11-05; First posted 2015-11-25 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Random Urine and 24 hour Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Prospective Blood Draw — This is prospective collection blood and urine study. This is not a treatment trial or device trial.

SUMMARY:
The study objectives are described below:

1. Obtain matched serum, plasma [(K2 EDTA, Sodium Heparin (NaH), Lithium Heparin (LiH)] and urine specimens collected from a minimum of 50 healthy subjects. Specimens will be used to determine a reference range for C-peptide and insulin assays, used as an aid in the assessment of C-peptide and insulin in adults.
2. Obtain serum and urine specimens collected from a minimum of an additional 200 healthy subjects. Specimens will be used to determine a reference range for C-peptide and insulin assays, used as an aid in the assessment of C-peptide and insulin in adults.
3. To store any remaining specimens for use in future assay development and to evaluate as yet undetermined assays for the development of IVDs, including additional C-peptide or insulin assays.

DETAILED DESCRIPTION:
The primary object of this study is to obtain a series of blood and urine specimens from women and men who are healthy with no history of abnormal blood sugar levels. The specimens will be used to evaluate new C-peptide and insulin assays (tests). Participants are being asked to voluntarily take part in this study because they are a healthy individual without a history of abnormal blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age ≥ 18 years
* Fasting for 12 hours prior to blood draw and random urine collection
* Able to understand and willing to provide informed consent
* Normal HbA1c (e.g. less than 5.7%) and glucose (e.g. less than 100 mg/dL) levels

Exclusion Criteria:

* Males and females, age <18 years
* Has a current diagnosis of any clinically significant cardiac, respiratory, neurological, immunological, hematological, liver disease, renal disease, gastrointestinal (GI) disorder, including any history of hyper- or hypothyroid, peptic or gastric ulcers or GI bleeding, or any other condition which, in the opinion of the investigator, would deem the subject unhealthy and therefore, ineligible.
* Has a history of any clinically significant cardiac, respiratory, neurological, immunological, hematological, liver disease, renal disease, gastrointestinal (GI) disorder, including any history of hyper- or hypothyroid, peptic or gastric ulcers or GI bleeding, or any other condition which, in the opinion of the investigator, is unstable at the time of enrollment.
* Current diagnosis or prior history of any type of diabetes including gestational diabetes.
* Currently taking or history of insulin therapy for any disease.
* Elevated HbA1c level (e.g. greater than 5.7%)
* Elevated glucose level (e.g. greater than or equal to 100 mg/dL)
* Is receiving systemic chemotherapy or radiation treatment, has an active malignancy of any type, or has been diagnosed with cancer within 5 years before screening other than basal or squamous cell skin cancers or in-situ cervical cancer.
* History of seizures
* Diagnosed with an infectious disease including any sexually transmitted diseases.
* Diagnosed with HIV/AIDS or ever tested positive for HIV.
* History of hepatitis
* Subject that has had sexual contact with a person who has hepatitis within the last 12 months.
* Pregnancy or lactation
* Non-fasting for 12 hours prior to blood and random urine collection.
* Hemolytic blood specimen
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 250 subjects will be enrolled in this study. Healthy women and men greater than or equal to 18 years of age having donated a single blood draw, a random urine specimen, and a 24-hour urine collection specimen will be eligible.
  Each site will evaluate and select patients for enrollment using the inclusion and exclusion criteria listed below. Study subjects should be selected from all available patients at the site. Each patient may be entered into the study only once.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Measure C-peptide and Insulin in Healthy Individuals | 10 months
  250 healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Diana Dickson, Study Director — Fujirebio Diagnostics, Inc.
Locations (1):
- Fundamental Research LLC, Gulf Shores, Alabama, United States